CLINICAL TRIAL: NCT01909037
Title: Exploratory Non Comparative Study to Evaluate the Efficacy of Highly Bioavailable Curcumin (Flexofytol) in Patients With Knee Osteoarthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tilman S.A. (Industry)
Collaborators: Bioxtract SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILFLEXFY 002
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-07

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; curcumin; biomarker; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

ARMS (1):
- Flexofytol (bio-optimized curcumin) (Experimental)
  Interventions: Dietary Supplement: Flexofytol (bio-optimized curcumin)

INTERVENTIONS:
Dietary Supplement: Flexofytol (bio-optimized curcumin) — 2x3 caps/day (before breakfast and in the evening) for 3 months

SUMMARY:
The purpose of this study is to evaluate the efficacy of bio-optimized curcumin(Flexofytol) during a 90-days period in knee ostearthritis patients on the serum levels of specific biomarkers of osteoarthritis and on the evaluation of pain.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 80 years of age
* Internal femorotibial gonarthrosis responding to the clinical and radiological criteria of ACR
* Symptomatic knee for more than 6 months
* Mean knee pain on the last 24 hours of at least 40 mm on VAS
* Kellgren & Laurence grade II to III
* Patients able to avoid NSAIDs and analgesics during the study
* Patients having signed informed consent
* Patients able to follow the study instructions

Exclusion Criteria:

* Related to the osteoarthritis pathology:

  * Osteoarthritis linked to a metabolic arthropathy
  * Predominant associated symptomatic femoropatellar osteoarthritis
  * Chondromatosis or villonodular synovitis of the knee
  * Recent trauma (< 1 month) of the knee responsible for the pain
  * Inflammatory flare
  * Pathology potentially interfering with the evaluation (metabolic inflammatory arthropathy, rheumatoid arthritis, lower limb radiculalgia, arthritis...
  * Paget disease
  * Homolateral coxarthrosis
  * Articular Prosthesis
  * Knee joint effusion
* Related to previous and associated treatments:

  * Corticosteroids injection in the previous month, whatever the joint concerned,
  * Hyaluronan injection in the evaluated knee during the previous 6 months,
  * NSAID or analgesics in the 72 hours prior to inclusion
  * No modification of Slow-acting drugs for OA and/or dietary supplements taken within less than 6 months prior to the study(ex: chondroitin sulfate, diacerein, soy and avocado unsaponifiables, oxaceprol, granions de cuivre, glucosamine, phytotherapy for OA, homeopathy for OA...),
  * Anticoagulant (coumarinic) treatment and heparin
  * General corticotherapy,
  * Contraindication to paracetamol.
* Related to associated pathologies:

  * Patient suffering from serious associated illness (liver failure, kidney failure, non-controlled cardiovascular diseases...)
* Related to patients:

  * Pregnant or breastfeeding women
  * Pre-menopausal women with no contraception
  * Patients unable to write
  * Patients enrolled in a clinical trial in the previous 3 months
  * Patients under juristic protection or under guardianship.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serum levels of biomarkers of cartilage metabolism and inflammation | 84 days
  Change from baseline of serum levels of biomarkers

SECONDARY OUTCOMES:
Pain and the global patient assessment of disease activity using a Visual Analog Scale (VAS) | 84 days
  Change from baseline of the mean pain over the last 24 hours and of the global assessment of disease activity by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Castermans, MD, Principal Investigator — Citadelle Hospital of Liege; Yvan Dierckxsens, Study Director — Tilman S.A.
Locations (1):
- Citadelle Hospital, Liège, Belgium

REFERENCES:
- [Derived] Henrotin Y, Gharbi M, Dierckxsens Y, Priem F, Marty M, Seidel L, Albert A, Heuse E, Bonnet V, Castermans C. Decrease of a specific biomarker of collagen degradation in osteoarthritis, Coll2-1, by treatment with highly bioavailable curcumin during an exploratory clinical trial. BMC Complement Altern Med. 2014 May 17;14:159. doi: 10.1186/1472-6882-14-159. PMID 24886572